CLINICAL TRIAL: NCT05261503
Title: Investigation of the Effectiveness of Environmental Enrichment-Based Intervention in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Cagla Sirma, PT, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EE Intervention in Preterm
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Preterm; Motor; Development, Infant; Therapy
Keywords: Preterm; Infant; Enriched Environment; Sensory; Motor; Development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homeostasis-Enrichment-Plasticity (Experimental): HEP group will receive an environmental enrichment-based intervention.
  Interventions: Other: HEP
- Traditional Physical Therapy (Experimental): TPT group will receive traditional physiotherapy intervention.
  Interventions: Other: Traditional Phsical Therapy

INTERVENTIONS:
Other: HEP — The Homeostasis-Enrichment-Plasticity (HEP) intervention group will receive 45 minutes of face-to-face environmental enrichment-based intervention one day per week and online home support once a week for 12 weeks.
  Arms: Homeostasis-Enrichment-Plasticity
Other: Traditional Phsical Therapy — The Traditional Physical Therapy group will receive a 45-minute intervention, two days a week for 12 weeks.
  Arms: Traditional Physical Therapy

SUMMARY:
The aim of this study is to investigate the effectiveness the HEP (Homeostasis-Enrichment-Plasticity) approach, which based upon the principles of enriched environment (EE) and ecological theories of development on preterm infants with developmental delay risk.

Thirty-two preterm infants aged 4-10 months will be randomly divided into 2 groups as the HEP intervention group and the Traditional Physical Therapy (TPT) group.

EE-based intervention will be applied to the HEP intervention group, and traditional physiotherapy will be applied to the TPT group for 12 weeks (24 sessions).

The demographic information of the participants will be recorded. The motor and sensory functions of the infants will be evaluated with, the Peabody Developmental Motor Scales (PDMS-2) and the Test of Sensory Functions in Infants™ (TSFI™), respectively. Additionally, the anxiety status of the parents will be evaluated with the Beck Anxiety Inventory (BAI). All evaluations will be done twice, at the end and at the beginning of 12 weeks.

DETAILED DESCRIPTION:
Premature birth is defined by WHO (World Health Organization) as all births occurring before 37 weeks of gestation. The global preterm birth rate for 2014 is estimated at 10.6% (9%-12%), equating to an estimated 14.84 million (12.65 million-16.73 million) live preterm births in 2014.

Preterm birth results in significant healthcare utilization and costs. Families of preterm infants often experience significant psychological and significant psychological and financial difficulties. Preterm infants have an increased risk for social, cognitive, language, sensory processing and motor skill disorders. There are different early intervention methods for preterm infants, and enriched environment (EE)-based intervention is one of the current intervention methods that have been used recently. There are studies showing that EE-based interventions have neurobehavioral benefits and positively affect brain functions and motor development.

There are a limited number of studies on EE-based early intervention methods in the literature, and these studies were conducted in different age and diagnosis groups by applying different intervention methods. Therefore, more studies are needed on this subject.

In this study, it was aimed to contribute to the literature in this field and to investigate the effectiveness of an EE-based intervention on the sensory and motor functions of preterm infants and the emotional state of the family.

ELIGIBILITY:
Inclusion Criteria:

* To be in corrected age between 4 and 10 months
* To being born 33 weeks and 6 days of gestation and before,
* To absence of any systemic disease, congenital anomaly,
* The family's volunteer to participate regularly in the study process.
* Having abnormal or suspect results on the Denver Developmental Screening Test II

Exclusion Criteria:

* To be born at or after 34 weeks of gestational age
* To having experienced intraventricular bleeding (Grade III and IV),
* To having major vision or hearing problems
* To having medical conditions that prevent active participation in the study (such as oxygen dependence)
* To participate in other experimental rehabilitation studies.

Ages: 4 Months to 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Motor Skills PDMS-2 Peabody Developmental Motor Scales 2nd Edition | 12 weeks
  The Peabody Developmental Motor Scales 2nd Edition (PDMS-2):
  PDMS-2 evaluates fine and gross motor skills of children from birth to six years of age relative to their peers. There are four subtests on gross motor skills (Reflexes, stationary performances, locomotion, object manipulation) and two subtests on fine motor skills (Grasping, visual-motor integration).
  In the test, the skills to be assessed are listed in chronological order. The test starts at the child's age-appropriate beginner level (the level at which he gets 2 points on three items in a row) and ends when the child scores 0 on each of the three items in a row.
  Each item is scored as 0 (does not show performance criteria), 1 (shows some of the performance criteria), 2 (shows performance criteria) according to the child's performance, and the total score for each section is calculated at the end of the test.
Sensory Function | 12 weeks
  Test of Sensory Functions in Infants™ (TSFI™):
  TSFI consists of 5 subtests and 24 items. The application time is approximately 20 minutes.
  In the subtests of the test, reactivity to tactile deep pressure, adaptive motor functions, visual-tactile integration, ocular-motor control, and reactivity to vestibular stimulation are evaluated and all items are scored.
  The infant is evaluated as normal, at-risk, or deficient in terms of sensory processing according to the total score he/she gets. A higher score indicates better sensory processing.

SECONDARY OUTCOMES:
Mental Health | 12 weeks
  Beck Anxiety Inventory (BAI):
  The Beck Anxiety Inventory (BAI) consists of 21 self-reported items that question physical and cognitive anxiety symptoms such as hot flashes, fear of something bad happening to oneself, heart palpitations, irritability, fear of drowning, and sweating not related to heat.
  The individual scores from 0 to 3 how intensely they have experienced these symptoms during the past week. The total score may range from 0 and 63: 0-7 points indicate minimal anxiety, 8-15 points indicate mild anxiety, 16-25 points indicate moderate anxiety, and 26-63 points indicate severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Aymen Balıkçı, Asst. Prof., Study Director — Fenerbahce University; Gamze Çağla Sırma, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)